CLINICAL TRIAL: NCT04397809
Title: Utility of CD64 and TLR2 Assays to Diagnose Acute Pulmonary Exacerbations in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14BGF-10
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Pulmonary Exacerbation (APE): Those subjects presenting with APE will be treated with at least two pathogen specific I.V. antibiotics, as dictated by their treating physician and compliant with standard guidelines for care of an APE.
- Baseline Health: Those subjects presenting at baseline health will be identified by their treating physician as such and will not be starting on any treatments for APE.

SUMMARY:
Cystic fibrosis (CF) is the most common inherited disease in the western world. On a yearly basis, 56% of CF patients, or nearly 17,000 individuals in the US, suffer from acute pulmonary exacerbations (APE). The purpose of this study is to test a candidate assay for its ability to diagnose APE, the most important disease event in CF. While previous studies have been able to identify biomarkers of CF prognosis and risk stratification, three markers have demonstrated characteristics ideal for APE diagnosis: CD64, TLR2, and GILT. CD64 is a cellular receptor, expressed on numerous cells of the immune system, whose role is to bind antibodies which are attached to infected cells or pathogens. TLR2 plays a major role in early host-microbial interactions. GILT has been shown to be more precise in targeting immune responses against antigens and influences T lymphocyte response. This study looks to identify the differences in the expression of neutrophil CD64 and CD4+ T cell TLR2 and GILT between acute illness and baseline health as a sensitive marker of acute pulmonary exacerbation so that it may facilitate rapid hematologic diagnosis of the condition. The study also looks to compare sensitivity and specificity of the assays above to standard measures, such as health related quality of life scores (CFQ-R), loss of lung function, white blood cell counts and CRP, for diagnosing acute exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF.
* Age 18 years old or greater.
* Presentation at baseline health OR at the start of treatment for a pulmonary exacerbation of CF.
* Ability to perform reproducible Pulmonary Function Tests
* Ability to produce sputum.
* Willingness to complete a health-related quality of life questionnaire
* Willingness to comply with study procedure and provide written consent.

Exclusion Criteria:

• Presence of a condition or abnormality that, in the opinion of the Principal Investigator (PI), would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CF patients aged 18 years or older at the time of an acute pulmonary exacerbation or at baseline health who are followed by the Adult CF Program at National Jewish Health will be eligible to enroll in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Difference in neutrophil CD64 expression | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  The primary outcome measure is the difference in expression of neutrophil CD64 as measured by flow cytometry from circulating blood between the two groups (APE and baseline).
Difference in CD4+ T cell TLR2 expression | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  The primary outcome measure is the difference in expression of CD4+ T cell TLR2 as measured by flow cytometry from circulating blood between the two groups (APE and baseline).
Difference in GILT expression | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  The primary outcome measure is the difference in expression of GILT as measured by flow cytometry from circulating blood between the two groups (APE and baseline).

SECONDARY OUTCOMES:
Correlation of primary outcome measurements with lung function tests | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  A secondary outcome measure is the correlation of the differences in expression of neutrophil CD64, CD4+ T cell TLR2, and GILT with changes in FEV1 as measured by spirometry.
Correlation of primary outcome measurements with C-Reactive Protein | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  A secondary outcome measure is the correlation of the differences in expression of neutrophil CD64, CD4+ T cell TLR2, and GILT with differences in C-Reactive Protein (CRP)
Correlation of primary outcome measurements with total white blood cell counts | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  A secondary outcome measure is the correlation of the differences in expression of neutrophil CD64, CD4+ T cell TLR2, and GILT with differences in total white blood cell counts (WBC).
Correlation of primary outcome measurements with sputum inflammatory markers | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  A secondary outcome measure is the correlation of the differences in expression of neutrophil CD64, CD4+ T cell TLR2, and GILT with differences in sputum inflammatory markers as measured by sputum neutrophil counts and neutrophil elastase expression.
Correlation of primary outcome measurements with phagocytosis | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  A secondary outcome measure is the correlation of the differences in expression of neutrophil CD64, CD4+ T cell TLR2, and GILT with differences in the percentage of phagocytosis by isolated neutrophils.
Correlation of primary outcome measurements with quality of life questionnaire score | Within 24 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation or at Baseline health
  A secondary outcome measure is the correlation of the differences in expression of neutrophil CD64, CD4+ T cell TLR2, and GILT with differences in patient reported health related quality of life scores as measured by the Cystic Fibrosis Questionnaire-Revised (CFQ-R).

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No